CLINICAL TRIAL: NCT00339482
Title: Prospective Studies of Diabetes Mellitus and Its Complications in the Gila River Indian Community
Brief Title: Prospective Studies of the Natural History of Diabetes Mellitus and Its Complications in the Gila River Indian Community
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 9999760256; OH76-DK-0256
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: AMERICAN INDIAN; Diabetes; Renal Diseases; Cardiovascular Disease; Natural History
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Kidney Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- American Indians: Residents of the Gila River Indian Community

SUMMARY:
This project is a continuation of an extensive longitudinal population-based epidemiological investigation of the etiology and determinants of type 2 diabetes (and its complications) and formerly arthritis. The original baseline observations were made on the residents of the Gila Indian Reservation, predominantly Pima Indians, in 1965. We attempt to reexamine the population at two-yearly intervals, and have continued to recruit new respondents who, because of age and residence or familial relationships, become eligible for entry into the project. Eligible persons receive a battery of standardized examinations related to diabetes and its complications at two-yearly intervals, including a glucose tolerance test, biochemical determinations, such as serum cholesterol and creatinine, insulin, etc., a physical examination, and in those aged 15 years and above, retinal photographs, and an electrocardiogram. Persons known to have diabetes will be asked to undergo the examination at annual intervals to enable more complete and accurate documentation of their health status and to identify the development and progression of complications of the disease.

The data collected have been used to describe the natural history and determinants of diabetes and its complications, to investigate factors relating to the etiology of these diseases and investigate the genetics of diabetes, its complications and other phenotypes. In addition, the project serves to identify subjects with specific characteristics for the clinical research projects carried out by the Obesity and Diabetes Clinical Research Section and the Diabetes Epidemiology and Clinical Research Section fo the Branch.

DETAILED DESCRIPTION:
This project is a continuation of an extensive longitudinal population-based epidemiological investigation of the etiology and determinants of type 2 diabetes (and its complications) and formerly arthritis. The original baseline observations were made on the residents of the Gila Indian Reservation, predominantly Pima Indians, in 1965. We attempt to reexamine the population at two-yearly intervals, and have continued to recruit new respondents who, because of age and residence or familial relationships, become eligible for entry into the project. Eligible persons receive a battery of standardized examinations related to diabetes and its complications at two-yearly intervals, including a glucose tolerance test, biochemical determinations, such as serum cholesterol and creatinine, insulin, etc., a physical examination, and in those aged 15 years and above, retinal photographs, and an electrocardiogram. Persons known to have diabetes will be asked to undergo the examination at annual intervals to enable more complete and accurate documentation of their health status and to identify the development and progression of complications of the disease.

The data collected have been used to describe the natural history and determinants of diabetes and its complications, to investigate factors relating to the etiology of these diseases and investigate the genetics of diabetes, its complications and other phenotypes. In addition, the project serves to identify subjects with specific characteristics for the clinical research projects carried out by the Obesity and Diabetes Clinical Research Section and the Diabetes Epidemiology and Clinical Research Section of the Branch.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study population is all persons aged 5 years and over residing on the Gila River Indian Reservation in Arizona. The vast majority of the eligible subjects are American Indians and there are similar numbers of males and females in the population. The study population was chosen because our previous work has shown that this population has the highest prevalence of Type 2 diabetes in the world. There are small numbers of other racial groups in the selected population who are also eligible to participate in the study. They are mainly members of the families in the community and therefore by participating they can contribute valuable research information to the study. All persons resident in the community aged 5 years and over are invited to participate in the study at two-yearly intervals. In addition, other tribal members and selected family members such as first or second degree relatives of the study population who reside, or have moved off the Reservation, are also eligible to participate.

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons aged 5 years and over residing in districts 1-5 of the Gila River Indian Community in Arizona.
Sampling Method: Non-Probability Sample
Enrollment: 12647 (Actual)
Dates: Start 1976-09-03 (Actual)

PRIMARY OUTCOMES:
To investigate the determinants of type 2 diabetes and its complications. | indefinite
  Development of diabetes and related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Hanson, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolford JK, Bogardus C, Prochazka M. Genome-wide scan for CAG/CTG repeat expansions in Pimas with early onset of type 2 diabetes mellitus. Mol Genet Metab. 1999 Jan;66(1):62-7. doi: 10.1006/mgme.1998.2775. PMID 9973549
- [Background] Lindsay RS, Dabelea D, Roumain J, Hanson RL, Bennett PH, Knowler WC. Type 2 diabetes and low birth weight: the role of paternal inheritance in the association of low birth weight and diabetes. Diabetes. 2000 Mar;49(3):445-9. doi: 10.2337/diabetes.49.3.445. PMID 10868967
- [Background] Silver K, Walston J, Yang Y, Pratley R, Ravussin E, Raben N, Shuldiner AR. Molecular scanning of the beta-3-adrenergic receptor gene in Pima Indians and Caucasians. Diabetes Metab Res Rev. 1999 May-Jun;15(3):175-80. doi: 10.1002/(sici)1520-7560(199905/06)15:33.0.co;2-y. PMID 10441039
- [Derived] Aydin BN, Stinson EJ, Hanson RL, Looker HC, Cabeza De Baca T, Krakoff J, Chang DC. Hepatic Insulin Resistance Increases Risk of Gallstone Disease in Indigenous Americans in the Southwestern United States. Clin Transl Gastroenterol. 2024 Nov 1;15(11):e00763. doi: 10.14309/ctg.0000000000000763. PMID 39166750
- [Derived] Mitchell CM, Stinson EJ, Chang DC, Krakoff J. A mixed meal tolerance test predicts onset of type 2 diabetes in Southwestern Indigenous adults. Nutr Diabetes. 2024 Jul 10;14(1):50. doi: 10.1038/s41387-024-00269-3. PMID 38987291
- [Derived] Stinson EJ, Mitchell CM, Looker HC, Krakoff J, Chang DC. Higher glucose and insulin responses to a mixed meal are associated with increased risk of diabetic retinopathy in Indigenous Americans. J Endocrinol Invest. 2024 Mar;47(3):699-707. doi: 10.1007/s40618-023-02187-0. Epub 2023 Sep 9. PMID 37684485
- [Derived] Shah MH, Piaggi P, Looker HC, Paddock E, Krakoff J, Chang DC. Lower insulin clearance is associated with increased risk of type 2 diabetes in Native Americans. Diabetologia. 2021 Apr;64(4):914-922. doi: 10.1007/s00125-020-05348-5. Epub 2021 Jan 6. PMID 33404681
- [Derived] Hohenadel MG, Baier LJ, Piaggi P, Muller YL, Hanson RL, Krakoff J, Thearle MS. The impact of genetic variants on BMI increase during childhood versus adulthood. Int J Obes (Lond). 2016 Aug;40(8):1301-9. doi: 10.1038/ijo.2016.53. Epub 2016 Apr 14. PMID 27076275
- [Derived] Hohenadel MG, Thearle MS, Grice BA, Huang H, Dai MH, Tao YX, Hunter LA, Palaguachi GI, Mou Z, Kim RC, Tsang MM, Haack K, Voruganti VS, Cole SA, Butte NF, Comuzzie AG, Muller YL, Baier LJ, Krakoff J, Knowler WC, Yanovski JA, Han JC. Brain-derived neurotrophic factor in human subjects with function-altering melanocortin-4 receptor variants. Int J Obes (Lond). 2014 Aug;38(8):1068-74. doi: 10.1038/ijo.2013.221. Epub 2013 Nov 26. PMID 24276017